CLINICAL TRIAL: NCT04196426
Title: Nutrition Education Intervention to Promote Dietary Calcium Intake Among Vietnamese Women Aged 30-65 Years in Rural Areas in Hanoi, Vietnam
Brief Title: Nutrition Education to Promote Calcium Intake Among 30-65 Year-old Women in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Hanoi University of Pharmacy (Unknown); Vietnam National Institute of Nutrition (Unknown)
Responsible Party: Principal Investigator, Bong, PhD Candidate, Texas Tech University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB2019-22
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Osteoporosis
Keywords: nutrition education; nutrition intervention; calcium intake; calcium-rich foods
MeSH Terms: conditions — Osteoporosis | interventions — Calcium

STUDY DESIGN:
Intervention Model Description: Three communities receive the nutrition intervention while three other communities do not. After 1 month, the first 3 communities do not receive the intervention while the later 3 communities receive the same nutrition intervention. Baseline, post intervention data are collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nutrition education group (Experimental): The nutrition education group receive the intervention first, which include 2 nutrition lessons about osteoporosis and calcium and calcium rich foods. The 2 lessons are delivered in one week for 2 hours each lesson. After this week, participants in the intervention group receive handouts about osteoporosis and calcium once a week for a period of 4 weeks.
  Interventions: Behavioral: Nutrition education intervention about osteoporosis and calcium
- delayed nutrition education group (Active Comparator): After the intervention group finish their intervention (5 weeks period), post data collection will be administered in both nutrition education and delayed nutrition education group. After this post data collection, the delayed nutrition education group receive the same intervention.
  Interventions: Behavioral: Nutrition education intervention about osteoporosis and calcium

INTERVENTIONS:
Behavioral: Nutrition education intervention about osteoporosis and calcium — The intervention is designed and developed based on the Intervention Mapping Process and the Health Belief Model. Topics of the intervention include: the importance of osteoporosis and risk factors, role of calcium in bone health and controlling the disease, calcium recommendations and sources, role of vitamin D and physical activity in calcium absorption and bone health, and how to identify calcium-rich foods in the locality and prepare meals with local calcium-rich foods. A recipe booklet containing recipes using local calcium-rich foods will be given to the participants after the end of the two nutrition lessons. Interactive activities are incorporated in each lesson to encourage the participation of participants.

SUMMARY:
Osteoporosis is an important public health problem in Vietnam, with one in ten Vietnamese women suffering from it. There is enough evidence demonstrating that low calcium intake is one of the risk factors for osteoporosis among Asian women in general and Vietnamese women in specific. It is reported that the intake of calcium among Vietnamese women is under 400 mg/day, which is less than the daily recommendation of 1,000 mg/day by the Vietnam National Institute of Nutrition, even though calcium-rich foods are largely available in Vietnam. Therefore, the purpose of this study is to promote dietary calcium intake among Vietnamese women aged 30-65 years through implementing a nutrition education intervention.

DETAILED DESCRIPTION:
Vietnamese women aged 30-65 years without medical problems that could interfere with the calcium consumption, such as kidney stone, kidney and liver diseases. The women will be excluded if they are blinded, deaf, or have general learning disability.

Outcomes of the study are dietary calcium intake, calcium knowledge, and osteoporosis health belief. A quantitative questionnaire is being used to collect these data.

ELIGIBILITY:
Inclusion Criteria:

* women aged 30 to 65 years

Exclusion Criteria:

* have medical conditions that can interfere with calcium intake, such as physician-diagnosed kidney stone, kidney and liver diseases, etc.
* blind, deaf, and have general learning disability

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Dietary calcium intake | 5 weeks
  The dietary calcium intake (mg/day) will be assessed using a food frequency questionnaire, which consisted of 36 food items contributing to the total calcium intake. The total calcium intake of each participant will be the sum of calcium intake from all food items in the food frequency questionnaire.

SECONDARY OUTCOMES:
Nutrition knowledge related to osteoporosis and calcium | 5 weeks
  The nutrition knowledge related to osteoporosis and calcium will be collected using a questionnaire that participants can answer by pencil. The knowledge included 11 question items. Participants received 1 point if answering correctly and 0 point if answering incorrectly. Total knowledge score ranged from 0 (minimum) to 11 points (maximum).
Osteoporosis health beliefs | 5 weeks
  Osteoporosis health beliefs will be collected using an osteoporosis health belief likert scale. The scale consisted of 6 subscales, including perceived susceptibility, perceived severity, perceived benefits, perceived barriers, health motivation, and self-efficacy. Each sub-scale of the health beliefs scale has 6 statements with 5 answering options, from "strongly disagree" (coded as 1) to "strongly agree" (coded as 5). Possible scores for each sub scale ranged from 6-30, with higher score indicating higher perception.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Murimi, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Preventive Medical Centers, Thach That, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared to other researchers. Any report that is generated will be based on aggregated data and will never identify individual responses.